CLINICAL TRIAL: NCT02697305
Title: Effect of Intravenously and Orally Administered Branched Chain Amino Acids on Incretin Response
Brief Title: Incretin Effects of Branched Chain Amino Acids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, MUDr. Radka Straková, MD, Charles University, Czech Republic
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IGA NT 14416 - 2
Record Dates: First submitted 2016-02-27; First posted 2016-03-03 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Glucose Metabolism Disorders
Keywords: Insulin response; Incretin effect; GLP-1; GIP; Valine; Leucine; Isoleucine; Branched chain amino acids
MeSH Terms: conditions — Glucose Metabolism Disorders | interventions — Methylcellulose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- IV BCAA test (Experimental): IV application of BCAA solution
  Interventions: Dietary Supplement: IV BCAA
- ORAL BCAA test (Experimental): At once oral ingestion of BCAA capsules
  Interventions: Dietary Supplement: ORAL BCAA
- ORAL PLACEBO test (Placebo Comparator): At once oral ingestion of placebo capsules
  Interventions: Other: ORAL Placebo

INTERVENTIONS:
Dietary Supplement: IV BCAA — in total dose of 0,4 g/kg in a 2 h intravenous infusion
  Other Names: Nutramin VLI 3%, Fresenius Kabi, KGaA, Germany
  Arms: IV BCAA test
Dietary Supplement: ORAL BCAA — single dose of 0.4g/kg administered over 30s washed down with 500mL of tap water
  Other Names: BCAA capsules, Reflex Nutrition, UK, Brighton
  Arms: ORAL BCAA test
Other: ORAL Placebo — single dose of 0.4 g/kg administered over 30 s washed down with 500mL of tap water
  Other Names: methylcellulose, University Hospital Inst. Pharmacy prepared
  Arms: ORAL PLACEBO test

SUMMARY:
Branched chain amino acids (BCAA) are known to exert insulinogenic effect. Whether this effect is mediated by incretins (GLP-1, GIP) is not known. The aim of the study was to show incretin effect of BCAA, i.e. whether the oral administration of BCAA elicits higher insulin and incretin response when compared with IV route of the same dose of BCAA. Eighteen healthy, male subjects participated in three tests: IV application of BCAA solution (30.7±1.1 g of BCAA, IV BCAA) second was oral ingestion of BCAA capsules in the same dose (ORAL BCAA) and third experiment was oral placebo (PLACEBO). Glucose, insulin, GLP-1, GIP, valine, leucine and isoleucine levels were measured at time interval for up to 4 h.

DETAILED DESCRIPTION:
Study protocols: Three tests were conducted on a different occasion (at least 7 days in between). First test (IV BCAA test) comprised of IV application of BCAA solution (Nutramin VLI 3%, Fresenius Kabi, KGaA, Germany; Leucine 43%, Isoleucine 24%, Valine 33%) in total dose of 0,4 g/kg in a 2 h infusion (mean solution volume 1023±34.6mL, mean total dose of BCAA 30.7±1.1g) to respect maximum recommended infusion rate. Second test (ORAL BCAA test) comprised of at once oral ingestion of BCAA capsules (BCAA capsules, Reflex Nutrition, UK, Brighton; Leucine 50%, Isoleucine 25%, Valine 25%) in a single dose of 0.4g/kg (mean total dose of BCAA 30.7±1.1 g) administered over 30s, washed down with 500mL of tap water. Third test (ORAL PLACEBO test) comprised of at once oral ingestion of placebo capsules (methylcellulose, University hospital institution pharmacy prepared) in a single dose of 0.4 g/kg administered over 30 s, washed down with 500 mL of tap water. The content of placebo capsules was weighted and packed identically with BCAA capsules. Nor participants nor the staff administering capsules and carrying out the protocol did not know about capsules content so that randomized double-blinded settings could have been maintained.

Blood analysis: Basal peripheral venous blood was drawn from each subject after 12 h of fasting (-15 min) and then at time 0, 15, 30, 45, 60, 90, 120, 150, 180, 210, 240 min throughout the intervention. Plasma was immediately separated and all samples were frozen at -80 °C until analysis were performed. For GLP-1 and GIP analysis BD P800 Blood Collection System was used with coat developed to preserve metabolic peptides in blood (cocktail of proteases, esterase and DPP-IV inhibitors, anticoagulant 3,6 mg di-potassium ethylenediaminetetraacetic acid (K2EDTA), Becton, Dickinson and Co., New Jersey, USA).

Parameters of glucose homeostasis were assessed: plasma glucose using hexokinase reaction (Konelab Glucose analyzer, Thermo Fisher Scientific, Oy., Finland) and serum insulin using solid phase competitive chemiluminescent enzyme immunoassay (Immulite 2000, Siemens A.G., Germany).

Commercially available ELISA kits were used for GLP-1 and GIP analysis: for GLP-1 Immuno-Biological Laboratories (Immuno-Biological Laboratories, Gunma, Japan) and for GIP Millipore (EMD Millipore Corporation, Bilerica, MA, USA).

Serum levels of BCAAs were determined by method of capillary electrophoresis (CE) with contactless conductivity detection, which has been already described in details [18]. Shortly: CE measurements were carried out using HP3DCE system (Agilent Technologies, Waldbronn, Germany) equipped with a built-in contactless conductivity detector. Separation took place in a fused-silica capillary (31.4 cm in total length, 14.7 cm to detector, 25 μm inside diameter, 363 μm outside diameter, Composite Metal Services, UK) at the controlled temperature of 25 °C. The inner surface of the capillary is covered using INST coating solution (Biotaq, U.S.A.) to prevent electro-osmotic flow before its first use [19]. The CE separation is performed in an optimized background electrolyte with composition 3.2 mol/l acetic acid in 20% v/v methanol, pH 2.0. The achieved separation time was 125 s at electric field intensity of 0.96 kV/cm and simultaneous application of a hydrodynamic pressure of 50 mbar. The separation efficiency in blood serum equaled 461,000 plates/m for valine and isoleucine, and 455,000 plates/m for leucine; the detection limits are equal to 0.4 µM for all three amino acids. The relative standard deviation values for repeatability of the migration time equaled 0.1% for measurements during a single day and 0.3% for measurements on different days; the relative standard deviation values for repeatability of the peak areas equaled 2.3 - 2.6% for measurements during a single day and 2.7 - 4.6% for measurements on different days. Blood samples were collected in test tubes containing ethylenediaminetetraacetic acid (EDTA). The obtained serum samples were stored in a freezer at -20 °C until the analysis. Prior to the analysis, the unfrozen serum samples were deproteinized by mixing 250 µl of serum with 750 µL of acetonitrile. Deproteinization was performed in an Eppendorf tube after shaking for 30s. Then the serum samples were centrifuged at an acceleration of 4 g for 45 s; 800 µL of the obtained supernatant were taken for CE analysis.

Statistical analysis: Data are presented in text, tables and figures as means ± standard error of the mean (SEM) and values of p<0.05 were considered statistically significant. Secretion responses for insulin, GIP, GLP-1, valine, leucine and isoleucine were calculated for each subject as incremental areas under the curve (iAUC). iAUCs calculation allow for different individual baseline values. iAUCs were calculated using the trapezoid model, from 0-240 min for glucose, insulin and BCAA and 0-120 for GLP-1 and GIP. All individual values below the baseline were excluded and each subject in respective study was their own reference. Secretion responses for glucose were calculated as decremental AUC (dAUC) as the response is predominantly negative. All individual values above the baseline were excluded in the case. Data for statistical comparison for iAUC and individual values were tested for normality and for normally distributed data, samples were compared using general linear model ANOVA with Bonferroni's multiple comparison to test the statistical significance of differences between groups. Repeated measures ANOVA test was used to assess time effect for every respective treatment. Mixed model ANOVA was used to assess treatment and time vs treatment effect. Differences between groups were identified using Bonferroni's multiple comparisons tests. GraphPad Prism, release 5.03 (GraphPad software, San Diego) was used to perform all statistical procedures.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers

Exclusion Criteria:

* age under 18 years, obesity, any chronic disease related to energy metabolism (particularly diabetes, thyreopathy, hypertension, dyslipidemia, atherosclerosis etc.), any chronic medication, smoking and regular alcohol consumption

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2014-09; Primary Completion 2015-05 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of GLP-1 and GIP | 0-120 min after administration
  At time 0, 15, 30, 45, 60, 90, 120 min serum levels of GLP-1 and GIP in peripheral blood samples were detected using commercially available ELISA kits

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of BCAA | 0-240 min after administration
  at time 0, 15, 30, 45, 60, 90, 120, 150, 180, 210, 240 min serum levels of BCAAs in peripheral blood samples were determined by method of capillary electrophoresis (CE) with contactless conductivity detection
Area under the plasma concentration versus time curve (AUC) of insulin | 0-240 min after administration
  at time 0, 15, 30, 45, 60, 90, 120, 150, 180, 210, 240 min serum levels of insulin in peripheral blood samples using solid phase competitive chemiluminescent enzyme immunoassay were detected
Area under the plasma concentration versus time curve (AUC) of glucose | 0-240 min after administration
  at time 0, 15, 30, 45, 60, 90, 120, 150, 180, 210, 240 min serum levels of glucose in peripheral blood samples using using hexokinase reaction were detected

CONTACTS AND LOCATIONS:
Overall Officials: Michal Anděl, Prof., MD, Principal Investigator — 3rd Faculty of Medicine, Charles University in Prague
Locations (1):
- Centre for Research on Diabetes, Metabolism and Nutrition, 3rd Faculty of Medicine, Charles University in Prague, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Berger S, Vongaraya N. Insulin response to ingested protein in diabetes. Diabetes. 1966 May;15(5):303-6. doi: 10.2337/diab.15.5.303. No abstract available. PMID 5936455
- [Background] Floyd JC Jr, Fajans SS, Conn JW, Knopf RF, Rull J. Stimulation of insulin secretion by amino acids. J Clin Invest. 1966 Sep;45(9):1487-502. doi: 10.1172/JCI105456. No abstract available. PMID 5919350
- [Background] Gannon MC, Nuttall FQ. Amino acid ingestion and glucose metabolism--a review. IUBMB Life. 2010 Sep;62(9):660-8. doi: 10.1002/iub.375. PMID 20882645
- [Background] Nilsson M, Stenberg M, Frid AH, Holst JJ, Bjorck IM. Glycemia and insulinemia in healthy subjects after lactose-equivalent meals of milk and other food proteins: the role of plasma amino acids and incretins. Am J Clin Nutr. 2004 Nov;80(5):1246-53. doi: 10.1093/ajcn/80.5.1246. PMID 15531672
- [Background] Frid AH, Nilsson M, Holst JJ, Bjorck IM. Effect of whey on blood glucose and insulin responses to composite breakfast and lunch meals in type 2 diabetic subjects. Am J Clin Nutr. 2005 Jul;82(1):69-75. doi: 10.1093/ajcn.82.1.69. PMID 16002802
- [Background] Pal S, Ellis V. The acute effects of four protein meals on insulin, glucose, appetite and energy intake in lean men. Br J Nutr. 2010 Oct;104(8):1241-8. doi: 10.1017/S0007114510001911. Epub 2010 May 11. PMID 20456814
- [Background] Layman DK. The role of leucine in weight loss diets and glucose homeostasis. J Nutr. 2003 Jan;133(1):261S-267S. doi: 10.1093/jn/133.1.261S. PMID 12514305
- [Background] Calbet JA, MacLean DA. Plasma glucagon and insulin responses depend on the rate of appearance of amino acids after ingestion of different protein solutions in humans. J Nutr. 2002 Aug;132(8):2174-82. doi: 10.1093/jn/132.8.2174. PMID 12163658
- [Background] Nilsson M, Holst JJ, Bjorck IM. Metabolic effects of amino acid mixtures and whey protein in healthy subjects: studies using glucose-equivalent drinks. Am J Clin Nutr. 2007 Apr;85(4):996-1004. doi: 10.1093/ajcn/85.4.996. PMID 17413098
- [Background] Wahren J, Felig P, Hagenfeldt L. Effect of protein ingestion on splanchnic and leg metabolism in normal man and in patients with diabetes mellitus. J Clin Invest. 1976 Apr;57(4):987-99. doi: 10.1172/JCI108375. PMID 947963
- [Background] Yang J, Chi Y, Burkhardt BR, Guan Y, Wolf BA. Leucine metabolism in regulation of insulin secretion from pancreatic beta cells. Nutr Rev. 2010 May;68(5):270-9. doi: 10.1111/j.1753-4887.2010.00282.x. PMID 20500788
- [Background] Raptis S, Dollinger HC, Schroder KE, Schleyer M, Rothenbuchner G, Pfeiffer EF. Differences in insulin, growth hormone and pancreatic enzyme secretion after intravenous and intraduodenal administration of mixed amino acids in man. N Engl J Med. 1973 Jun 7;288(23):1199-202. doi: 10.1056/NEJM197306072882302. No abstract available. PMID 4700552
- [Background] ELRICK H, STIMMLER L, HLAD CJ Jr, ARAI Y. PLASMA INSULIN RESPONSE TO ORAL AND INTRAVENOUS GLUCOSE ADMINISTRATION. J Clin Endocrinol Metab. 1964 Oct;24:1076-82. doi: 10.1210/jcem-24-10-1076. No abstract available. PMID 14228531
- [Background] Nauck MA, Homberger E, Siegel EG, Allen RC, Eaton RP, Ebert R, Creutzfeldt W. Incretin effects of increasing glucose loads in man calculated from venous insulin and C-peptide responses. J Clin Endocrinol Metab. 1986 Aug;63(2):492-8. doi: 10.1210/jcem-63-2-492. PMID 3522621
- [Background] Gunnerud U, Holst JJ, Ostman E, Bjorck I. The glycemic, insulinemic and plasma amino acid responses to equi-carbohydrate milk meals, a pilot- study of bovine and human milk. Nutr J. 2012 Oct 12;11:83. doi: 10.1186/1475-2891-11-83. PMID 23057765
- [Background] Salehi A, Gunnerud U, Muhammed SJ, Ostman E, Holst JJ, Bjorck I, Rorsman P. The insulinogenic effect of whey protein is partially mediated by a direct effect of amino acids and GIP on beta-cells. Nutr Metab (Lond). 2012 May 30;9(1):48. doi: 10.1186/1743-7075-9-48. PMID 22647249
- [Background] Chen Q, Reimer RA. Dairy protein and leucine alter GLP-1 release and mRNA of genes involved in intestinal lipid metabolism in vitro. Nutrition. 2009 Mar;25(3):340-9. doi: 10.1016/j.nut.2008.08.012. Epub 2008 Nov 26. PMID 19036562
- [Background] Tuma P, Gojda J. Rapid determination of branched chain amino acids in human blood plasma by pressure-assisted capillary electrophoresis with contactless conductivity detection. Electrophoresis. 2015 Aug;36(16):1969-75. doi: 10.1002/elps.201400585. Epub 2015 Apr 8. PMID 25639649
- [Background] Tuma P. Rapid determination of globin chains in red blood cells by capillary electrophoresis using INSTCoated fused-silica capillary. J Sep Sci. 2014 Apr;37(8):1026-32. doi: 10.1002/jssc.201400044. Epub 2014 Mar 13. PMID 24677638
- [Background] Rocha DM, Faloona GR, Unger RH. Glucagon-stimulating activity of 20 amino acids in dogs. J Clin Invest. 1972 Sep;51(9):2346-51. doi: 10.1172/JCI107046. PMID 4639019
- [Background] Pedroso JA, Zampieri TT, Donato J Jr. Reviewing the Effects of L-Leucine Supplementation in the Regulation of Food Intake, Energy Balance, and Glucose Homeostasis. Nutrients. 2015 May 22;7(5):3914-37. doi: 10.3390/nu7053914. PMID 26007339
- [Background] Palmer JP, Benson JW, Walter RM, Ensinck JW. Arginine-stimulated acute phase of insulin and glucagon secretion in diabetic subjects. J Clin Invest. 1976 Sep;58(3):565-70. doi: 10.1172/JCI108502. PMID 783201
- [Background] Vahl TP, Drazen DL, Seeley RJ, D'Alessio DA, Woods SC. Meal-anticipatory glucagon-like peptide-1 secretion in rats. Endocrinology. 2010 Feb;151(2):569-75. doi: 10.1210/en.2009-1002. Epub 2009 Nov 13. PMID 19915164
- [Background] Marina AS, Kutina AV, Shakhmatova EI, Balbotkina EV, Natochin YV. Stimulation of glucagon-like peptide-1 secretion by water loading in human. Dokl Biol Sci. 2014 Nov;459:323-5. doi: 10.1134/S0012496614060027. Epub 2015 Jan 6. No abstract available. PMID 25560206
- [Background] Yang J, Wong RK, Park M, Wu J, Cook JR, York DA, Deng S, Markmann J, Naji A, Wolf BA, Gao Z. Leucine regulation of glucokinase and ATP synthase sensitizes glucose-induced insulin secretion in pancreatic beta-cells. Diabetes. 2006 Jan;55(1):193-201. PMID 16380493
- [Background] van Loon LJ, Kruijshoop M, Menheere PP, Wagenmakers AJ, Saris WH, Keizer HA. Amino acid ingestion strongly enhances insulin secretion in patients with long-term type 2 diabetes. Diabetes Care. 2003 Mar;26(3):625-30. doi: 10.2337/diacare.26.3.625. PMID 12610012
- [Background] Solerte SB, Fioravanti M, Locatelli E, Bonacasa R, Zamboni M, Basso C, Mazzoleni A, Mansi V, Geroutis N, Gazzaruso C. Improvement of blood glucose control and insulin sensitivity during a long-term (60 weeks) randomized study with amino acid dietary supplements in elderly subjects with type 2 diabetes mellitus. Am J Cardiol. 2008 Jun 2;101(11A):82E-88E. doi: 10.1016/j.amjcard.2008.03.006. PMID 18514633
- [Derived] Gojda J, Strakova R, Plihalova A, Tuma P, Potockova J, Polak J, Andel M. Increased Incretin But Not Insulin Response after Oral versus Intravenous Branched Chain Amino Acids. Ann Nutr Metab. 2017;70(4):293-302. doi: 10.1159/000475604. Epub 2017 Jun 9. PMID 28595189